CLINICAL TRIAL: NCT01480726
Title: Endoscopic Versus Open Vein Harvest in Coronary Artery Bypass Grafting. Clinical and CT-angiographic Long-term Result From a Randomized Study.
Brief Title: Long-term Results Following Endoscopic Vein Harvesting in Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Jan Jesper Andreasen, MD, PhD, Professor, MD, PhD, Aalborg University Hospital
Other Study IDs: N20110023
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2011-11

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open vein harvest: Conventional open vein harvest from the lower leg
  Interventions: Procedure: Surgery
- Endoscopic vein harvest: Endoscopic vein harvest from the calf
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery

SUMMARY:
Vena saphena magna is still frequently used as graft material in coronary artery bypass grating(CABG, and vein grafts can harvest with either the conventional open technique (Ovh = open vein harvesting), or with less invasive endoscopic techniques (EVH = Endoscopic vein harvesting). The endoscopic techniques have been shown to reduce the incidence of postoperative wound complications while patients are more satisfied with the cosmetic result of the operation on the leg.

Non-randomized studies have raised doubts about patency rates of the vein grafts following EVH compared to OVH, while other studies failed to detect any problems in relation to this. There are only very few data on long-term patency rates from randomized studies.

The purpose of this study is to investigate clinical outcome and patency rates of the vein grafts following either EVH and OVH in 132 patients who underwent CABG for 4-7 years ago as part of a randomized study investigation wound complications. A cost-effectiveness analysis will also be performed.

The hypothesis is: Patency rates following EVH are worse compared to OVH in CABG 4-7 years postoperatively.

DETAILED DESCRIPTION:
Background

Vena saphena magna is frequently used as graft material in coronary artery bypass grafting (CABG. Vein grafts can be harvested with conventional open technique (OVH = open vein harvesting), or with various endoscopic less invasive techniques (EVH = Endoscopic vein harvesting). The endoscopic techniques have been shown to reduce the incidence of postoperative wound complications and patients are more satisfied with the cosmetic surgery results.

Non-randomized trials, however, cast doubt on the patency rates of the vein grafts following EVH compared to OVH, while other studies including one randomized trial failed to detect any problems regarding this. There are no data regarding long-term patency rate following EVH.

It is therefore valuable to conduct a secondary follow-up among CABG patients who 4-7 years ago were included in a randomized trial focusing on wound complications from the leg. Although the study was not designed to evaluate the clinical results and patency rates of vein graft, such a study may still contribute with important knowledge because the results will come from a randomized patient cohorts, in contrast to results from most other studies.

Purpose

To investigate long-term patency rates (4-7 years) patency rates and clinical outcomes following EVH and OVH in first-time CABG.

We also want to perform a health economic analysis (cost-effectiveness analysis) to assess which of the two harvesting methods.

Hypotheses:

1. Patency rates following EVH are worse compared to OVH in CABG 4-7 years postoperatively.
2. EVH is associated with an increased incidence of recurrence of angina and the need for re-revascularization compared with OVH.
3. Although EVH immediately leads to higher direct costs compared with OVH, there is a health economic benefit of this method in the long run.

Methods:

This experiment consists of a follow-up among 129 of 132 former patients who underwent first-time CABG between April 2004 - June 2007 at Aalborg Hospital, Aarhus University Hospital, Denmark, comparing EVH and OVH. Register data will be collected and patient records will be reviewed. Surviving patients will be invited for a clinical evaluation. CT-angio in order to compare long-term patency rates of the vein grafts will be performed. Furthermore the incidence of recurrent angina, acute coronary syndrome, need for re-revascularization and cardiovascular death since the operation wil be evaluated.

All direct and indirect costs of the two methods of surgery and throughout the postoperative course until this study will be valued in order to perform a health economic analysis (cost-effectiveness analysis).

Subjects The age of the previous trial subjects was 65 years (range 43-90 years, at the time they were included in the previous study, and survivors will be 4-7 years old today.

It is expected that most of the surviving former patients will participate in the study.

Inclusion Criteria

All 129 former patients who were included in the initial trial may be included. Deceased patients are only included in the trial regarding registry data and medical records.

Exclusion criteria (in relation to the clinical examination):

Lack of consent. (Register Data for previous patients who did not give their informed consent for a clinical follow-up may be included in the study)

Exclusion criteria (in relation to CT-angio):

Former patients with at least one of the following exclusion criteria will not have a CT-angio performed:

p-creatinine> 120 micromol / l Estimated GFR (eGFR = estimated glomerular filtration rate) per 1.73 m2 <60 ml / min.

Atrial fibrillation Allergy to contrast media Pregnancy Breastfeeding Lack of consent

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the previous randomized study
* Informed consent from the patient

Exclusion Criteria:

* Survival until date of reexamination
* No informed consent
* CT scan of the heart will not be performed in patients with if: atrial fibrillation,p-creatinin >120 micromol/l, allergy to contrast, pregnancy, lactating.

Ages: 43 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 132 patients who underwent CABG 4-7 years ago. All patients participated in a randomized study focusing on wound complications from the leg following either open or endoscopic vein harvest.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Patency rates of vein grafts | 5-7 years postoperatively

SECONDARY OUTCOMES:
recurrence of angina pectoris | 5-7 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jan J. Andreasen, MD. PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark